CLINICAL TRIAL: NCT05197075
Title: A Study to Assess the Acceptability of the Darunavir/Cobicistat (DRV/COBI) Fixed-dose Combination (FDC) Tablet in Human Immunodeficiency Virus (HIV)-1 Infected Children Aged >=3 Years and Weighing >=15 kg to <25 kg
Brief Title: A Study to Assess the Acceptability of the Darunavir/Cobicistat (DRV/COBI) Fixed-dose Combination (FDC) Tablet in Human Immunodeficiency Virus (HIV)-1 Infected Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CR109146; 2021-000738-32 (EudraCT Number); TMC114FD1HTX1001 (Other: Janssen Research and Development, LLC)
Record Dates: First submitted 2022-01-17; First posted 2022-01-19 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Human Immunodeficiency Virus (HIV)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Darunavir/Cobicistat (DRV/COBI) Fixed Dose Combination (FDC) (Experimental): Participants will receive the DRV/COBI FDC tablet for oral use, dispersed in water on Day 1.
  Interventions: Drug: DRV/COBI FDC

INTERVENTIONS:
Drug: DRV/COBI FDC — DRV/COBI FDC tablet dispersed in water will be administered orally.
  Other Names: TMC114/JNJ-48763364

SUMMARY:
The purpose of the study is to assess the ability to swallow the Darunavir/Cobicistat (DRV/COBI) fixed dosed combination (FDC) tablet dispersed in water.

DETAILED DESCRIPTION:
Human immunodeficiency virus type 1 (HIV-1) infection is a life-threatening and serious disease that is of major public health interest around the world. Standard-of-care for the treatment of HIV infection involves the use of a combination of antiretroviral (ARV) drugs to suppress viral replication to below detectable limits, to increase CD4+ cell count, and to delay disease progression. Darunavir (DRV) is an inhibitor of the dimerization and of the catalytic activity of the HIV-1 protease. It selectively inhibits the cleavage of HIV encoded Gag-Pol polyproteins in virus infected cells, thereby preventing the formation of mature infectious virus particles. Cobicistat (COBI) is a mechanism-based inhibitor (MBI) of the cytochrome P450 (CYP)3A subfamily. Inhibition of CYP3A mediated metabolism by COBI enhances the systemic exposure of CYP3A substrates, such as DRV, where bioavailability is limited and half-life is shortened by CYP3A-dependent metabolism. DRV/COBI FDC tablet formulation would overcome the difficulties of pediatric participants (greater than or equal to [>=] 3 years and weighing >=15 kilograms [kg] to less than [<] 25 kg) might encounter in swallowing a whole or 2 halves of an oral, non-disintegrating tablet, hence helping children to better adhere to their HIV treatment. The study consists of a screening phase (up to 21 days) and an open-label administration phase of 1 day. Safety will be assessed by adverse events (AEs). The total duration of the study is up to 32 days.

ELIGIBILITY:
Inclusion Criteria

* Has documented chronic Human Immunodeficiency Virus (HIV-1) infection
* Must be on an allowed stable unchanged antiretroviral (ARV) regimen for at least 3 months prior to screening
* Has a documented plasma HIV-1 Ribonucleic acid (RNA) less than 400 copies/milliliters (mL) within 6 months prior to or at screening
* Must be in a condition that allows to perform the protocol-specified assessments and so must his/her caregiver, if applicable. If a participant and his or her caregiver have difficulties in completing the questionnaire, the study-site personnel may assist
* Body weight within greater than or equal to (>=) 15 kilograms (kg) to less than (<) 25 kg

Exclusion criteria

* Known allergies, hypersensitivity, or intolerance to Darunavir/Cobicistat (DRV/COBI) or any excipient of the study intervention
* Has taken any disallowed therapies
* Any active condition (example, active oral infection [candidiasis], significant physical or psychological disease or other findings during screening) that could prevent the participant from swallowing dispersions in water, or for which, in the opinion of the investigator, participation would not be in the best interest of the participant (example, compromise the well-being) or that could prevent, limit, or confound the protocol specified assessments and outcomes
* Active acquired immunodeficiency syndrome (AIDS)-defining illness at screening
* Has had any contact with severe acute respiratory syndrome coronavirus 2 (SARS CoV 2) positive or Coronavirus Disease 2019 (COVID-19) participants within the last 2 weeks prior to admission to the clinical research center

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2022-09-23 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Ability to Take the Darunavir/Cobicistat (DRV/COBI) Fixed Dosed Combination (FDC) Tablet Dispersed in Water as Reported by the Observer | Day 1
  The percentage of participants that is able to swallow the medication fully versus partially or not at all, based on the questionnaire for the observer will be reported.

SECONDARY OUTCOMES:
Ease of Swallowing of Tablet Dispersed in Water by the Participant | Day 1
  Ease of Swallowing of tablet dispersed in water by the participant will be assessed by using 5-point hedonic scale acceptability questionnaire to be completed by the participant indicating how difficult/easy it is to swallow the tablet dispersed in water (very difficult, difficult, ok, easy, and very easy).
Ease of Swallowing of Tablet Dispersed in Water by the Participant as Reported by the Caregiver | Day 1
  Ease of Swallowing of tablet dispersed in water by the participant will be assessed by using 5-point hedonic scale acceptability questionnaire to be completed by the caregiver on the basis of reaction/ facial expression of the participant, indicating how difficult/easy it is for the participant to swallow the tablet dispersed in water (very difficult, difficult, ok, easy, and very easy).
Palatability of the Tablet Dispersed in Water by the Participant | Day 1
  Palatability of tablet dispersed in water by the participant will be assessed by using 5-point hedonic scale acceptability questionnaire indicating the taste of the tablet dispersed in water (dislike very much, dislike a little, not sure, like a little, like a lot).
Palatability of the Tablet Dispersed in Water by the Participant as Reported by the Caregiver | Day 1
  Palatability of tablet dispersed in water by the participant will be assessed by using 5-point hedonic scale acceptability questionnaire to be completed by the caregiver on the basis of reaction/ facial expression of the participant, indicating how the participant like the taste of the tablet dispersed in water (dislike very much, dislike a little, not sure, like a little, like a lot).
Ease of Dispersion of the Tablet in the Water as Reported by the Caregiver | Day 1
  Ease of dispersion of the tablet in the water will be assessed by using 5-point hedonic scale acceptability questionnaire to be completed by the caregiver, indicating how difficult/easy it is to disperse the tablet in water (very difficult, difficult, ok, easy, and very easy).
Acceptability of Taking the Tablet Dispersed in Water Everyday by the Participant | Day 1
  Acceptability of taking the tablet dispersed in water everyday by the participant will be assessed by using 5-point hedonic scale acceptability questionnaire indicating how difficult/easy it is to take the tablet everyday (very difficult, difficult, ok, easy, and very easy).
Acceptability of Taking the Tablet Dispersed in Water Everyday by the Participant as Reported by the Caregiver | Day 1
  Acceptability of taking the tablet dispersed in water everyday by the participant will be assessed by using 5-point hedonic scale acceptability questionnaire to be completed by the caregiver, indicating how difficult/easy it is for the participant to take the tablet everyday (very difficult, difficult, ok, easy, and very easy).
Number of Participants with Adverse Event | Up to 32 days
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research and Development, LLC Clinical Trial, Study Director — Janssen Research and Development LLC
Locations (6):
- Emory University, Atlanta, Georgia, United States
- South Africa (2):
  - Rahima Moosa Mother and Child Hospital, University of Witwatersrand, Johannesburg
  - Global Clinical Trials PE, Pretoria
- Spain (3):
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Hosp. Clinico San Carlos, Madrid
  - Hosp. Univ. La Paz, Madrid

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency